CLINICAL TRIAL: NCT04683042
Title: Fibromyalgia TENS in Physical Therapy Study (TIPS): an Embedded Pragmatic Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kathleen Sluka (Other)
Responsible Party: Sponsor-Investigator, Kathleen Sluka, Kathleen A. Sluka, PhD, PT, FAPTA, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201909757; 1UG3AR076387-01 (NIH)
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia
Keywords: Transcutaneous Electrical Nerve Stimulation (TENS); chronic pain; fibromyalgia; movement pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study is a pragmatic clinical trial in outpatient PT practices utilizing cluster randomization by facility and facility size. Sites will be randomized to enroll all eligible and consented participants with FM to TENS with PT, or PT only (no TENS). We have identified 25-35 clinics across 6 healthcare systems in both rural and urban settings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TENS with PT (Active Comparator): TENS with PT group: The TENS with PT group will receive usual PT care and following enrollment, during the second PT visit, participants will receive TENS units and instruction on use of the TENS units. TENS will be applied to the upper and lower back with butterfly electrodes using the following parameters: mixed frequency (2-125Hz), strong but comfortable intensity, variable pulse duration from 100-250 microseconds. TENS to be applied when the patient is active and doing exercises at home and during PT sessions for 30 minutes at least 2 hours per day. The TENS with PT group will complete TENS use to the end of the study at 6 months.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS) with PT
- No TENS with PT (Other): The No TENS group will receive usual PT care until the primary endpoint timeframe of 60 days. After completion of the research homework at 60 days, TENS units will be mailed to the participants and a study team member will complete virtual TENS instruction. The no TENS group will complete TENS to the end of the study at 6 months.
  Interventions: Other: PT only

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) with PT — Use of TENS units along with routine PT therapy
  Arms: TENS with PT
Other: PT only — Routine PT therapy only
  Arms: No TENS with PT

SUMMARY:
The purpose of this study is to determine if addition of Transcutaneous Electrical Nerve Stimulation (TENS) to routine physical therapy improves movement-evoked pain in patients with fibromyalgia (FM).

The study will also determine if addition of TENS to routine physical therapy (PT) improves disease activity and symptoms, increases adherence to physical therapy, increases the likelihood of meeting patient specific functional goals, and reduces medication use.

DETAILED DESCRIPTION:
This study is a pragmatic clinical trial in outpatient PT practices utilizing cluster randomization by healthcare system and facility size. Sites will be randomized to enroll all eligible and consented participants with FM to TENS with PT, or PT only (no TENS). We are identifying 25-35 clinics across 6 healthcare systems in both rural and urban settings. We will enroll 450 patients that self report a clinician diagnosis of FM. At each site, TENS (or no TENS) will be applied during each visit along with individualized PT treatment specified by the physical therapist. Participants randomized to TENS intervention sites will receive TENS units and electrodes at baseline to be applied to the cervical and lumbar regions. Participants will take the units home and bring the units back to their PT clinic visits with instructions for use at home while active and during their exercises. The physical therapist at each clinic will complete routine documentation of treatment. In addition to the primary and secondary outcomes, Electronic Health Record data variables will be collected as exploratory outcomes. Variables including adherence to treatment will be extracted from each site's Electronic Health Record. Patient-reported assessments will be obtained from the participant's at home the day of their second PT visit (Baseline) and at 30, 60 (primary outcome), 90, and 180 days following enrollment. The primary and secondary outcome assessments will be comparing TENS and no TENS groups in terms of changes from baseline to 60 days.

Participants will be identified after they are referred for PT for treatment of primary fibromyalgia (FM) or chronic pain (pain lasting more than three months). At their first (intake) physical therapy visit, they will be provided information about the study that can be accessed on paper or on-line. They will perform an electronic screening form on the first visit if interested in participating. Participants will provide e-consent after eligibility is confirmed at the initial PT visit. At the second PT visit after e-consent is signed, participants will be provided instructions on logging onto REDCap for data capture and accessing the case report forms. Participants enrolled at a TENS site will then be instructed in use of TENS and the TENS unit with electrodes will be provided. Those participants enrolled at a no TENS site will skip the instruction in use of TENS but will then receive instructions along with the TENS units at day 65. Participants will be instructed to capture all baseline assessments at home before their next PT visit before and following their first TENS treatment (or no TENS) at home (day 1). At 30, 60, 90, and 180 days following enrollment, participants will complete the same assessments at home including pain ratings at rest and with movement along with questionnaires. The primary and secondary outcome assessments will be comparing TENS and no TENS groups in terms of changes from baseline to 60 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 until 99.
2. Clinician diagnosis of FM
3. Referred for land-based PT
4. Referred for treatment for FM or chronic pain (pain lasting more than 3 months)
5. Able to provide informed consent.
6. Fluent in reading English
7. Willing to use TENS

Exclusion Criteria:

1. Contraindications to TENS use including:

   1. Pacemaker, defibrillator, implanted neurostimulator or implanted device
   2. Epilepsy
   3. Currently pregnant or plan to become pregnant in the next 6 months
   4. Allergic reaction to patches with gel
   5. Current treatment for cancer
2. Currently enrolled in another pain control study
3. Use of TENS within the last 30 days
4. Clinically unstable medical or psychiatric issues

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Reduction of movement-evoked pain (0-10 Low to High scale) during the Sit and Stand Test | Research Homework before PT Visit 3 (Day 1), Day 60 +/- 5 days Home
  Numeric rating scale of 0-10 for reduction of movement-evoked pain measured by 11-point NRS from baseline to 60 days.

SECONDARY OUTCOMES:
Change in the resting pain score (0 - 10 Low to High scale) | Research Homework before PT Visit 3 (Day 1), Day 60 +/- 5 days Home
  The severity of pain will be measured on a 0 to 10 numeric rating scale where 0 is no-pain and 10 is worst pain imaginable.
Pain interference (BPI) (0-10 Low to High Scale) | Research Homework before PT Visit 3 (Day 1), Day 60 +/- 5 days Home
  11 items measuring pain severity and interference with daily activities on a 0-10 scale.
FM Disease activity (FIQR) (0-10 Low to High Scale) | Research Homework before PT Visit 3 (Day 1), Day 60 +/- 5 days Home
  21 items used to evaluate function, overall impact, and symptoms in patients with fibromyalgia.
Resting fatigue (NRS) (0-10 Low to High Scale) | Research Homework before PT Visit 3 (Day 1), Day 60 +/- 5 days Home
  The severity of fatigue will be measured with a 0 to 10 scale where 0 is no fatigue and 10 is worst fatigue imaginable.
Movement-evoked fatigue (NRS) (0-10 Low to High Scale) | Research Homework before PT Visit 3 (Day 1), Day 60 +/- 5 days Home
  Fatigue during a five times sit and stand test will be measured with a 0 to 10 numeric rating scale with 0 as no fatigue and 10 as the worst fatigue imaginable.
Multidimensional assessment of fatigue (MAF) (0-10 Low to High Scale) | Research Homework before PT Visit 3 (Day 1), Day 60 +/- 5 days Home
  16 items measuring fatigue according to four dimensions: degree and severity, distress that it causes, timing of fatigue, and impact on various activities of daily living.
Rapid assessment of physical activity (RAPA) (0-10 Low to High Scale) | Research Homework before PT Visit 3 (Day 1), Day 60 +/- 5 days Home
  9 items evaluating current level of physical activity.
Patient global impression of change (PGIC) (0-6 Scale) | Day 60 +/- 5 days Home
  Evaluates overall health status as perceived by the patient in a seven-point single-item scale ranging from 'very much worse' to 'very much improved'

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Sluka, PhD, PT, Principal Investigator — University of Iowa; Leslie Crofford, MD, Principal Investigator — Vanderbilt University; Dana Dailey, PhD, PT, Study Director — University of Iowa
Locations (6):
- United States (6):
  - University of Illinois at Chicago, Chicago, Illinois
  - Rock Valley Physical Therapy, Moline, Illinois
  - Kepros Physical Therapy and Performance, Cedar Rapids, Iowa
  - Genesis Physical Therapy, Davenport, Iowa
  - Big Stone Therapies (BST), Big Stone City, South Dakota
  - Advanced Physical Therapy Sport Medicine, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The current study is expected to generate patient-reported outcomes for individuals with fibromyalgia across a broad spectrum of domains, pain, fatigue, function, psychological factors, and quality of life. We will also collect some data from the electronic health record about number of physical therapy visits, Current Protocol Terminology (CPT) codes for treatments, and the patient-specific functional scale. In addition, we will have TENS usage data downloaded from the TENS devices that will show the number of minutes of TENS use and the number of 30 minute sessions completed. Data will be collected prior to the intervention (baseline data) and 30, 60, 90 and 180 days after enrollment.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Analysis datasets will be made available at the time of publication of the primary manuscript. Complete datasets and accompanying resources will be deposited to the designated NIH Helping to End Addiction Long-term initiative (HEAL) data repository after the completion of the primary aim manuscript.
Access Criteria: In accordance with NIH Collaboratory policies, we will prepare the primary analysis datasets (at a minimum) for submission to the Collaboratory Coordinating Center. In accordance with International Committee of Medical Journal Editors (ICMJE) policies, we will prepare the primary analysis datasets for review and reproducibility by peer-reviewed journals. We will prepare the final datasets and accompanying resource documents for final deposit to the designated NIH HEAL data repository.
  Publications will be made available to the public using open access publishing, so they become available immediately to the public. All publications will be accessible through PubMED, google scholar, and available to the public through open access.

REFERENCES:
- [Derived] Post AA, Dailey DL, Bayman EO, Chimenti RL, Costigan M, Franck C, Huff T, Johnson E, Koepp M, Lafontant DE, McCabe ME, Neill-Hudson T, Vance CGT, Van Gorp B, Zimmerman BM, Ecklund D, Crofford LJ, Sluka KA. The Fibromyalgia Transcutaneous Electrical Nerve Stimulation in Physical Therapy Study Protocol: A Multisite Embedded Pragmatic Trial. Phys Ther. 2022 Nov 6;102(11):pzac116. doi: 10.1093/ptj/pzac116. PMID 36036838

DOCUMENTS (3):
  • Study Protocol (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT04683042/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT04683042/SAP_001.pdf
  • Informed Consent Form (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT04683042/ICF_002.pdf